CLINICAL TRIAL: NCT05783960
Title: Multicenter External Validation of Clinical Prediction Tools for Estimating Salt and Potassium . Study UniverSel
Brief Title: External Validation of Clinical Prediction Tools for Estimating Salt and Potassium Intake in Nephrology Patients.
Acronym: UniverSel
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0239
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Diseases
Keywords: salt diet; potassium diet; prediction tools; Bayesian network; kidney disease; epidemiology
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- External validation a questionnaire: Questionnaire will be administrated to patient with chronic kidney diseases ti evaluated the consumption of salt and potassium intake. A Bayesian network and a multiple regression will be used to validated the questionary of 27 items
  Interventions: Other: administration questionary

INTERVENTIONS:
Other: administration questionary — Questionnaire will be compared to 24h sodium and potassium urinary excretion (reference). A Bayesian network and a multiple regression will be used to validate the questionary
  Other Names: administration questionary 27 items to evaluate the salt and potassium intake

SUMMARY:
There is no validated self-questionnaire to assess salt and potassium intake in nephrology patients.

Using Bayesian models, researchers developed clinical prediction tools to estimate salt and potassium intake in nephrology patients. These prediction tools performed well, with an accuracy of 89% for salt and 74% for potassium, and have undergone internal validation.

Currently, the investigators wish to conduct an external validation study of these clinical prediction tools using data from patients followed at 3 nephrologic centers to generalize the performance results of the tools.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* Consultant or inpatient in the nephrology department
* Having performed a 24-hour urinary assessment as part of his usual management with analysis of natriuresis and/or kaliuresis.

Exclusion Criteria:

* Patient having lost salt by vomiting, diarrhea and intense sweating (sport) in the week preceding the 24-hour urine collection.
* Person protected by the french law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of patients consulting or hospitalized in day hospital in the nephrology department of one of the three centers participating in the study: Hôpital Lyon Sud (Hospices Civils Lyon), AURAL (Association pour l'Utilisation du Rein Artificiel dans la région Lyonnaise) Lyon and Hôpitaux Universitaires de Bordeaux. It is therefore composed of patients suffering from different types of nephropathy (lithiasis, diabetes, hypertension, tubulo interstitial, glomerular, autosomal dominant polycystic or other) whatever the stage of their disease and of healthy volunteers (living donors).
Sampling Method: Non-Probability Sample
Enrollment: 629 (Actual)
Dates: Start 2023-07-16 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
External multicenter validation questionary | at inclusion
  comparison of answers to the questionnaire about salt and potassium diet with natriuresis and kaliuresis urinary excretion during 24 hours administrated in 3 centres in nephrology in France

CONTACTS AND LOCATIONS:
Overall Officials: Jean Pierre Fauvel, Principal Investigator — Service Nephrologie, Hôpital Edouard Herriot
Locations (5):
- France (5):
  - Service de néphrologie Hôpitaux Universitaires de Strasbourg, Strasbourg, Alsace
  - AURAL, Lyon
  - Hopital Lyon SUD, Lyon
  - HÖPITAL bichat, Paris
  - CHU Rangueil, Toulouse